CLINICAL TRIAL: NCT06438003
Title: Improving Healthy Living Opportunities: Laurel HARVEST
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Makenzie Barr-Porter (Other)
Responsible Party: Sponsor-Investigator, Makenzie Barr-Porter, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 64602; 2022-68015-36497 (Other Grant/Funding Number: USDA NIFA)
Record Dates: First submitted 2024-05-24; First posted 2024-05-31 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Health Knowledge, Attitudes, Practice; Obesity
Keywords: Health Equity; Food Insecurity; Rural
MeSH Terms: conditions — Behavior; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laurel County (Experimental): Specialized services
  Interventions: Behavioral: Special Services
- Pike County (Active Comparator): Extension services as usual
  Interventions: Other: Services as Usual

INTERVENTIONS:
Behavioral: Special Services — Community members will complete data collection at the extension office or community partner location. Extension cooking classes and helping to make raised bed gardens along with other area happenings will be offered to participants throughout the year with check-ins and reminders. Data will be collected from study participants (regardless of the intervention decided) , at two time points, to include survey, dietary recall, and carotenoid scanner.
  Arms: Laurel County
Other: Services as Usual — Community members will receive extension services as usual with Data collection on participants at two time points to assess changes in rates of food insecurity, dietary quality, and overall health conditions.
  Arms: Pike County

SUMMARY:
The goal of this pre-post intervention study is to understand how community-engaged approaches to policy, systems, and environmental approaches can work to improve fruit and vegetable consumption and food security status among an Appalachian Kentucky community. The main approaches taken will be to employ a Community Advisory Board to define our target population of need, and appropriate intervention strategies. The investigators aim to understand if nutrition-based programming and food system approaches for lower-income, single-parent households, and multi-generational households can improve health. Participants will engage in annual data collection to assess dietary quality and food security status.

ELIGIBILITY:
Inclusion Criteria:

* Resident of Laurel of Pike County
* Over 18 years of age

Exclusion Criteria:

* Pregnancy
* Non-English speaking
* Plans to move out of the counties within the next three years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2023-01-27 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
change in food security | Baseline (year 1) and year 3
  Food Security Status will be measured at each time point by the 10-item United States Department of Agriculture (USDA) Household Food Security Module. The questionnaire includes ten questions pertaining to food security that were designed to assess an individual's ability to obtain food directly to ensure having enough healthy food to eat. The questions include items such as not having enough money to purchase food, inability to afford nutritious food, and skipping meals due to lack of sufficient money. Answer choices include often, sometimes, never, and don't know. Items will be scored Food security status is assigned as follows: raw score zero-High food security among adults, raw score 1-2-Marginal food security, raw score 3-5-Low food security, raw score 6-10-Very low food security. For some reporting purposes, the food security status of the first two categories in combination will be described as food secure and the latter two as food insecure.
change in total Healthy Eating Index scores | Baseline (year 1) and year 3
  The Healthy Eating Index is a measurement that can capture changes in the thirteen dietary components outlined in the Dietary Guidelines for Americans. A maximum score-5 or 10 points- can be reached for each dietary component, depending on the component. Points are awarded when the amounts consumed meets the standard for a particular dietary component. Amounts that do not meet the standard get fewer points, with zero being the minimum score, and the maximum total Healthy Eating Index score is 100.
Change in Food and Physical Activity Questionnaire (FPAQ) | Baseline (year 1) and year 3
  30 item questionnaire to collect self-reported behaviors pertaining to five domains: diet, physical activity, food safety, food security and food resource management. The response options for each question are based on a Likert scale. Each question is scored with higher scores indicating greater frequency of the behavior in question.
change in carotenoids | Baseline (year 1) and year 3
  the VEGGIE METER™ will be used to measure dermal carotenoids using non-invasive RS Spectroscopy. Carotenoids are a biological marker of fruit and vegetable consumption. This non-invasive measurement of dermal carotenoids has been validated against the standard of serum carotenoids in adults. To obtain the measurement, a subject places their pointer finger into the machine for 20 seconds while their finger is squeezed. Three replicates will be taken per person at 20 seconds per replicate. The VEGGIE METER™ scores dermal carotenoids on a scale of 0-850 with higher scores indicating higher intake.

CONTACTS AND LOCATIONS:
Overall Officials: Makenzie Barr-Porter, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/03/NCT06438003/ICF_000.pdf